CLINICAL TRIAL: NCT04355819
Title: Patient Centered Outcomes Among Patients With and Without Ventral Hernia
Brief Title: Patient Centered Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Julie Holihan, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-16-0698
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure before (Experimental): Patients will be told that a hernia was found on CT before the follow-up survey is administered.
  Interventions: Behavioral: Disclosure timing
- Disclosure after (Experimental): Patients will be told that a hernia was found on CT after the follow-up survey was administered.
  Interventions: Behavioral: Disclosure timing

INTERVENTIONS:
Behavioral: Disclosure timing — When patients are told that a hernia was present on the CT scan

SUMMARY:
Several questions exist when looking at ventral hernias:

1. what is the baseline quality of life and abdominal wall function among patients with or without a ventral hernia?
2. what is the clinical significance of a ventral hernia seen on radiography but not on clinical examination (e.g. occult hernia)?
3. what is the natural history of quality of life of patients with and without a ventral hernia?
4. what is the impact of disclosure of presence or absence of a ventral hernia on quality of life?

Answering these questions can provide valuable information on the impact of surgery with or without subsequent ventral hernia on a patient's abdominal wall function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Patients at LBJ Hospital
* Patients who received a CT of the abdomen

Exclusion Criteria:

* Children (under age 18 years old)
* Any patient in any vulnerable population (e.g pregnant women, prisoners, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Patient Centered Outcomes (PCO) | Consent to 1 year follow-up
  Difference in PCO from initial survey to follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Julie Holihan, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olavarria OA, Lyons NB, Bernardi K, Dhanani NH, Neela N, Arakelians A, Cohen BL, Mohebzad K, Coelho R, Holihan JL, Liang MK. Impact of disclosure of radiographic test results on quality of life among patients with hernias: a randomized controlled trial. Hernia. 2024 Apr;28(2):411-418. doi: 10.1007/s10029-023-02824-w. Epub 2023 Jun 27. PMID 37369887